CLINICAL TRIAL: NCT04359797
Title: Pragmatic Trial Exploring Impact of Patient Positioning in the Management of Patients Infected With COVID-19: Supine vs. Prone
Brief Title: COVID-19 Patient Positioning Pragmatic Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Todd Rice, MD, MSc, Associate Professor, Department of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200727
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Results first posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic controlled clinical trial with parallel group assignment.
Who Masked: Outcomes Assessor
Masking Description: Patients and providers will necessarily be unblinded, but outcomes will be analyzed by a blind assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to this arm will remain in their natural choice of position, which is anticipated to favor a supine, semi-recumbent position.
  Interventions: Other: Usual Care
- Prone (Active Comparator): Participants randomized to this arm will be encouraged to lay in a completely prone position for as much time as is tolerable during hospitalization.
  Interventions: Other: Prone

INTERVENTIONS:
Other: Prone — Provider-recommended guidance on prone positioning of patients
  Other Names: Proning
  Arms: Prone
Other: Usual Care — No provider-recommendation, patients will remain in their natural choice of position
  Arms: Usual Care

SUMMARY:
This study aims to determine if provider-recommended guidance on supine (on back) vs. prone (on stomach) positioning of patients testing positive for COVID-19 requiring supplemental oxygen, but not yet mechanically ventilated, improves outcomes in the inpatient setting. This study will be performed as a pragmatic clinical trial.

DETAILED DESCRIPTION:
Disease Progression and Timing of Intervention The intervention described herein focuses on adjustment of patient positioning aimed at improving gas exchange and lung function in patients harboring COVID-19. This intervention will target the inpatient setting generally.

Scientific/Clinical Rationale for Approach Since emergence of the novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) now designated coronavirus disease 2019 (COVID-19), one in six affected patients becomes seriously ill. The lung appears to be the most susceptible target organ, with a large swath of symptomatic patients struggling with mild upper respiratory tract illness and severe viral pneumonia resulting in respiratory failure. This respiratory failure is often fatal, with one study showing 28% non-survivors having experienced respiratory failure. Moreover, 81-97% of patients requiring mechanical ventilation do not survive.

Like its interaction with Severe Acute Respiratory Syndrome (SARS-CoV), angiotensin converting enzyme 2 (ACE2) is the functional receptor for COVID-19. Viral adherence to host-cell membrane associated ACE2 facilitates the proximity required for viral "spike" mediated genetic material injection. In COVID-19, this spike is 10-20 times more likely to bind ACE2 than SARS. ACE2 is expressed in 0.64% of all human lung cells, with 83% of those cells being alveolar epithelial type II. In addition, gene ontology enrichment analysis showed that the ACE2-expressing alveolar epithelial type II have high levels of multiple viral process-related genes, including regulatory genes for viral processes, viral life cycle, viral assembly, and viral genome replication, suggesting that the ACE2-expressing alveolar epithelial type II cells facilitate coronaviral replication in the lung. Thus, these cells likely serve as a ready reservoir for viral invasion. Perhaps more importantly, alveolar type II cells function to generate and recycle surfactant essential to respiratory activity. Surfactant defends against alveolar collapse at low lung volume and protects the lung from injuries/infections caused by inhaled particles and micro-organisms. In COVID-19, if these vital cells are being destroyed, alveolar failure may ensue with severe lung impairment. Thus, interventions that are aimed at improving pressure normalization and alveolar protection may be beneficial in these patients.

Prone positioning (PP) has long been used to combat hypoxemia in acute respiratory distress syndrome (ARDS). Improvements in gas exchange result from improved alveolar ventilation and blood flow redistribution with enhanced perfusion following. PP reduces lung over inflation and bolsters alveolar recruitment. PP also promotes uniformity of vertical pleural pressure gradients resulting in more uniform alveolar size. Considering these physiologic factors together, the investigators hypothesize PP serves to balance stress and strain within the lungs of non-critically ill patients with COVID-19 leading to improved outcomes compared to traditional supine positioning.

Prior Research Supporting the Positioning Model:

Multiple studies have been conducted that support the use of PP as a proactive treatment to combat hypoxemia in ARDS. Each year, approximately 170,000 people are diagnosed with ARDS, and those diagnosed face mortality rates between 25% and 40%. The use of PP stretches back to the 1970s, as providers began to search for ways to ameliorate ARDS symptomatology and reduce the then even higher levels of mortality associated with it. Following initial reports that PP significantly improved oxygenation in 70-80% of patients with ARDS, it was adopted as a standard treatment option. Initially, randomized clinical trials struggled to replicate these findings, citing multiple limitations to study enrollment and treatment standardization that made ascertaining conclusive results difficult. Only as RCT construction has been refined to accommodate for these limitations have the benefits of PP been more clearly demonstrated.

These beneficial effects have been recently upheld by the landmark PROSEVA study, a multicenter, prospective, randomized, controlled trial, that randomly assigned 466 patients with severe ARDS to undergo prone-positioning sessions of at least 16 hours or to be left in the supine position. Their results demonstrated a significant improvement in both 28- and 90-day mortality rates: "the 28-day mortality was 16.0% in the prone group and 32.8% in the supine group (P<0.001). The hazard ratio for death with prone positioning was 0.39 (95% confidence interval [CI], 0.25 to 0.63). Unadjusted 90-day mortality was 23.6% in the prone group versus 41.0% in the supine group (P<0.001), with a hazard ratio of 0.44 (95% CI, 0.29 to 0.67)".

Per these positive findings, PP has been consistently shown to be an effective mechanism to increase oxygenation in patients with ARDS when implemented under the following conditions: early enlisting of treatment and its consistent maintenance for at least 16 hours per day, and with concurrent use of lung-protective therapies. Translating these findings towards treatment of COVID-19 positive patients seems promising given the similarity of manifested symptoms and complications.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll all patients admitted to VUMC who test positive for COVID-19 and require supplemental oxygen, but are not yet mechanically ventilated.

Exclusion Criteria:

* Patients admitted on mechanical ventilation will be excluded from enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Highland Park, Illinois
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Q&A on coronaviruses (COVID-19) [Internet]. [cited 2020 Mar 24];Available from: https://www.who.int/news-room/q-a-detail/q-a-coronaviruses
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Feb 24 SS| NR| CN|, 2020. Study of 72,000 COVID-19 patients finds 2.3% death rate [Internet]. CIDRAP. [cited 2020 Mar 24];Available from: http://www.cidrap.umn.edu/news-perspective/2020/02/study-72000-covid-19-patients-finds-23-death-rate
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Wrapp D, Wang N, Corbett KS, Goldsmith JA, Hsieh CL, Abiona O, Graham BS, McLellan JS. Cryo-EM structure of the 2019-nCoV spike in the prefusion conformation. Science. 2020 Mar 13;367(6483):1260-1263. doi: 10.1126/science.abb2507. Epub 2020 Feb 19. PMID 32075877
- [Background] Zhao Y, Zhao Z, Wang Y, Zhou Y, Ma Y, Zuo W. Single-cell RNA expression profiling of ACE2, the putative receptor of Wuhan 2019-nCov. bioRxiv 2020;2020.01.26.919985.
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Background] Andreeva AV, Kutuzov MA, Voyno-Yasenetskaya TA. Regulation of surfactant secretion in alveolar type II cells. Am J Physiol Lung Cell Mol Physiol. 2007 Aug;293(2):L259-71. doi: 10.1152/ajplung.00112.2007. Epub 2007 May 11. PMID 17496061
- [Background] Johnson NJ, Luks AM, Glenny RW. Gas Exchange in the Prone Posture. Respir Care. 2017 Aug;62(8):1097-1110. doi: 10.4187/respcare.05512. Epub 2017 May 30. PMID 28559471
- [Background] Galiatsou E, Kostanti E, Svarna E, Kitsakos A, Koulouras V, Efremidis SC, Nakos G. Prone position augments recruitment and prevents alveolar overinflation in acute lung injury. Am J Respir Crit Care Med. 2006 Jul 15;174(2):187-97. doi: 10.1164/rccm.200506-899OC. Epub 2006 Apr 27. PMID 16645177
- [Background] Kallet RH. A Comprehensive Review of Prone Position in ARDS. Respir Care. 2015 Nov;60(11):1660-87. doi: 10.4187/respcare.04271. PMID 26493592
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Pickham D, Berte N, Pihulic M, Valdez A, Mayer B, Desai M. Effect of a wearable patient sensor on care delivery for preventing pressure injuries in acutely ill adults: A pragmatic randomized clinical trial (LS-HAPI study). Int J Nurs Stud. 2018 Apr;80:12-19. doi: 10.1016/j.ijnurstu.2017.12.012. Epub 2017 Dec 30. PMID 29331656
- [Background] Schutt SC, Tarver C, Pezzani M. Pilot study: Assessing the effect of continual position monitoring technology on compliance with patient turning protocols. Nurs Open. 2017 Oct 26;5(1):21-28. doi: 10.1002/nop2.105. eCollection 2018 Jan. PMID 29344391
- [Derived] Qian ET, Gatto CL, Amusina O, Dear ML, Hiser W, Buie R, Kripalani S, Harrell FE Jr, Freundlich RE, Gao Y, Gong W, Hennessy C, Grooms J, Mattingly M, Bellam SK, Burke J, Zakaria A, Vasilevskis EE, Billings FT 4th, Pulley JM, Bernard GR, Lindsell CJ, Rice TW; Vanderbilt Learning Healthcare System Platform Investigators. Assessment of Awake Prone Positioning in Hospitalized Adults With COVID-19: A Nonrandomized Controlled Trial. JAMA Intern Med. 2022 Jun 1;182(6):612-621. doi: 10.1001/jamainternmed.2022.1070. PMID 35435937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Prone
Started | 243 | 258
Completed | 243 | 258
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Prone | Total
Number analyzed (Participants) | 243 | 258 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (15.2) | 61.6 (15.4) | 61.0 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 112 | 217
  Male | 138 | 146 | 284
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 162 | 154 | 316
  Race: Black or African American | 43 | 56 | 99
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 6 | 8 | 14
  Race: Other race | 26 | 30 | 56
  Race: Unknown race | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic/Latinx | 204 | 213 | 417
  Ethnicity: Hispanic/Latinx | 33 | 33 | 66
  Ethnicity: Unknown ethnicity | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  United States | 243 | 258 | 501

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized on the Modified WHO Ordinal Scale by the Highest Level of Support on Day 5
Description: The highest level of support on the 5th day after enrollment according to the following scale adjusted for patient status at enrollment according to the same scale and ranked by mean FIO2 within each category, as appropriate.
  * Death
  * ECMO
  * Mechanical ventilation (ranked by mean FIO2)
  * Non-invasive ventilation such as BiPAP (ranked by mean FIO2)
  * High flow nasal cannula, e.g. Optiflow, Vapotherm or other similar device (titrated by FiO2%) (ranked by mean FIO2)
  * Standard nasal cannula (titrated by L/min up to 15 L/min) or face mask (ranked by mean FIO2)
  * Room air
Time Frame: 5 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Prone
Number analyzed (Participants) | 243 | 258
Participants
  Discharged | 109 | 99
  Room Air | 15 | 15
  Standard Nasal Cannula | 57 | 65
  High Flow Nasal Cannula | 16 | 16
  Non-invasive Ventilation | 26 | 24
  Mechanical Ventilation | 10 | 19
  ECMO | 1 | 1
  Death | 9 | 19

2. Secondary Outcome: FIO2
Description: For each day, the investigators will record the most intensive oxygen delivery mode and then, for that highest level of oxygen support device, the max FiO2 while exposed to that device.
Time Frame: First 5 days post-randomization
Measure: Mean (Standard Deviation); unit: percentage of inspired oxygen
Arm/Group | Usual Care | Prone
Number analyzed (Participants) | 243 | 258
percentage of inspired oxygen
  Day 1 | 40.4 (27.1) | 45.3 (29.1)
  Day 2 | 40.3 (28.2) | 44.0 (30.9)
  Day 3 | 39.3 (29.8) | 43.6 (32.1)
  Day 4 | 37.8 (30.2) | 42.7 (32.5)
  Day 5 | 37.1 (31.0) | 40.6 (32.0)

ADVERSE EVENTS:
Time Frame: 28 days
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Usual Care | Prone
All-Cause Mortality (participants affected / at risk) | 48/243 | 63/258
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/258
Other Adverse Events (participants affected / at risk) | 0/243 | 0/258

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04359797/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04359797/SAP_001.pdf